CLINICAL TRIAL: NCT04318483
Title: Clinical and Biological Description of an Atypical IgE-mediated Cow Milk Allergy (CMA) Form With Hands and Feet Angio-oedema From the Diagnosis to Its Spontaneous Evolution and Comparison to the Typical CMA Form Without Oedema of Extremities
Brief Title: Characteristic and Evolution of an Atypical IgE-mediated Cow Milk Allergy Form With Hands and Feet Angio-oedema
Acronym: IgE-CMA
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 19-HPNCL-04
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Angio-oedema of extremities: Patients who had revealed IgE-mediated cow milk allergy with hands and feet oedema
  Interventions: Other: survey
- Without angio-oedema of extremities: Patients who had revealed IgE-mediated cow milk allergy with hands and feet oedema
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — parents' telephone interview to collect medical history

SUMMARY:
Cow milk allergy is one of the most frequent food allergy among children. Cow milk protein's avoidance is needed until spontaneous recovery during the two first years of life. A atypical clinical form with angio-oedema of hands and feet which is associated with high rate of lactoserum's IgE might be a hope of an earlier recovery.

DETAILED DESCRIPTION:
Cow Milk allergy is one of the most frequent pediatric food allergy and occurs during the first months of life. It is due to an inappropriate reaction of immune system against the human body. Its treatment is the avoidance of the cow milk proteins. Its spontaneous recovery occurs mostly during the first years of life with the decreasing of the specific IgE and the clinical tolerance to cow milk proteins.

Two shorts cas reports (3 and 5 patients) have described a clinical form of IgE-mediated cow milk allergy with angio-oedema of hands and feet. This clinical form is associated with more increasing of specific IgE against lactoserum proteins than caseine's. However it has been showed that casein is a marker of cow milk allergy persistence. It might be possible that this atypical form of cow milk allergy progresses favorably towards a restoration of tolerance earlier than the clinical form without angio-oedema of the extremities

ELIGIBILITY:
Inclusion Criteria:

* Patients with a concordant history of IgE-mediated CMA (skin reaction within the next hours of cow milk proteins intake, regression of symptoms with avoidance of cow milk, +/- recurrence of identical symptoms when readministration)
* Patients with documented positive awareness markers (skin test and/or specific IgE > 0,1 kilo units of allergen-specific IgE per liter (kUA/l ))
* Patient followed at the pediatric allergology consultation at the Pediatric Hospitals of Nice

Exclusion Criteria:

* patients without IgE specific performed in the first month after the reaction
* patients who have had only 1 documented specific IgE test

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient followed at the pediatric allergology consultation at the Pediatric Hospitals of Nice
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
kinetics of specific IgE | at inclusion
  kinetic is defined by dosage of specific IgE (cow milk, caseine, whey proteins) from diagnostic from control to 7 months after

SECONDARY OUTCOMES:
comparison of specific IgE kinetics between case and control patient | at inclusion
  Respective evolution of the kinetics of specific IgE directed against whey proteins and casein between T0 and T1
Clinical characteristics of allergic reaction | at inclusion
  description of cow milk allergy : associated clinical signs, kinetics of appearance of clinical signs, kinetics of disappearance, treatment undertaken
Clinical characteristics of patients | at inclusion
  description of another allergy
Age of clinical tolerance | at inclusion
  age of clinical tolerance is defined by age of food reintroduction at home or at hospital